CLINICAL TRIAL: NCT01556724
Title: A Comparison of 0.1 and 0.2% Ropivacaine in Lumbar Plexus Catheters After Primary Total Hip Arthroplasty: a Comparison of Postoperative Analgesia and Motor Function.
Brief Title: A Comparison of Postoperative Analgesic Nerve Block Ropivacaine Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sylvia Wilson (Other)
Responsible Party: Sponsor-Investigator, Sylvia Wilson, Regional Anesthesia Fellow, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO09090339
Record Dates: First submitted 2012-03-06; First posted 2012-03-16 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Total Hip Arthroplasty; Postoperative Pain
Keywords: Peripheral nerve blocks; Ropivacaine concentrations in lumbar plexus catheters; Postoperative pain; Total hip replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.2% ropivacaine nerve block (standard of care) (Active Comparator): 0.2% ropivacaine in lumbar plexus nerve catheter infusions for postoperative analgesia
  Interventions: Drug: 0.1% or 0.2% ropivacaine nerve blocks
- 0.1% ropivacaine infusion in nerve block catheter (Experimental): 0.1% ropivacaine in lumbar plexus nerve catheter infusions
  Interventions: Drug: 0.1% or 0.2% ropivacaine nerve blocks

INTERVENTIONS:
Drug: 0.1% or 0.2% ropivacaine nerve blocks — Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuous lumbar plexus catheters will be removed on post operative day (POD) 2.
  Other Names: Naropin (ropivacaine hcl)

SUMMARY:
Peripheral nerve blocks are the standard of care for pain management after hip replacement surgery at UPMC Shadyside. This prospective, randomized study is intended to assess the effect of 0.1 versus 0.2% ropivacaine in lumbar plexus nerve catheter infusions after total hip arthroplasty. Ropivacaine peripheral nerve block infusions have been utilized as the standard of care at UPMC Shadyside for many years. Ropivacaine, a less potent left-isomer of bupivacaine, is often used in place of bupivacaine due to less motor blockade and less severe cardiovascular and central nervous system potential toxicity.

The primary goal of this study to examine the effect of a low concentration infusion of ropivacaine (0.1%) on postoperative analgesia (evaluated by opioid consumption after 36 hours) compared with the standard accepted concentration of 0.2% ropivacaine in lumbar plexus catheters after primary total hip arthroplasty. Secondary goals are to examine motor function, VAS scores and patient satisfaction with pain control in low concentration 0.1% ropivacaine compared with 0.2% ropivacaine lumbar plexus infusions upto 36 hours after primary total hip arthroplasty.

DETAILED DESCRIPTION:
Lumbar plexus catheters are the standard of care for postoperative pain management following total hip arthroplasty (THA) at UPMC Shadyside. The safety and efficacy of this technique has been demonstrated by multiple studies. Ropivacaine 0.2% was used for many years at UPMC Shadyside and throughout the UPMC system and this concentration of ropivacaine is the standard local anesthetic utilized by multiple other studies. However, this concentration of ropivacaine was later decreased to 0.1% in our institution in order to decrease patient's motor weakness and promote postoperative physical therapy. Patients were clinically observed to continue to have adequate postoperative analgesia while demonstrating improved motor function. A randomized, double blinded clinical trial has never compared 0.1 and 0.2% ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* American Society of Anesthesiologists physical status score I-III
* Scheduled for primary total hip arthroplasty at UPMC Shadyside Hospital in Pittsburgh, PA.
* No contraindications to peripheral nerve catheter placement
* Patients not expected to receive therapeutic anticoagulation in the postoperative period.
* No known drug allergies to study medications
* Patients willing to receive spinal anesthesia as operative anesthetic

Exclusion Criteria:

* Age under 18 years or older than 75 years.
* Any contraindication to a placement of continuous lumbar plexus peripheral nerve catheter.
* American Society of Anesthesiologist physical status IV or greater.
* Chronic painful conditions.
* Preoperative opioid tolerant use (opioid use for greater than 6 contiguous months before surgery).
* Coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively.
* Allergy to any of the drugs/agents used study protocol.
* Pregnancy
* Having an altered mental status (not oriented to place, person, or time)
* Any comorbid condition that, in the judgment of the consulting orthopedic surgeon or intraoperative anesthesiologist, would proscribe the patient from any aspect of the study.
* Patient refusal.
* Patient requiring postoperative management in the ICU
* Lumbar plexus catheter placed by loss of resistance technique.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, MD, Principal Investigator — University of Pittsburgh Medical Center; Jacques E Chelly, MD, PhD, MBA, Study Chair — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Siddiqui ZI, Cepeda MS, Denman W, Schumann R, Carr DB. Continuous lumbar plexus block provides improved analgesia with fewer side effects compared with systemic opioids after hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):393-8. doi: 10.1016/j.rapm.2007.04.008. PMID 17961837
- [Background] Marino J, Russo J, Kenny M, Herenstein R, Livote E, Chelly JE. Continuous lumbar plexus block for postoperative pain control after total hip arthroplasty. A randomized controlled trial. J Bone Joint Surg Am. 2009 Jan;91(1):29-37. doi: 10.2106/JBJS.H.00079. PMID 19122076
- [Background] Zink W, Graf BM. Local anesthetic myotoxicity. Reg Anesth Pain Med. 2004 Jul-Aug;29(4):333-40. doi: 10.1016/j.rapm.2004.02.008. PMID 15305253
- [Background] Leone S, Di Cianni S, Casati A, Fanelli G. Pharmacology, toxicology, and clinical use of new long acting local anesthetics, ropivacaine and levobupivacaine. Acta Biomed. 2008 Aug;79(2):92-105. PMID 18788503
- [Background] Paauwe JJ, Thomassen BJ, Weterings J, van Rossum E, Ausems ME. Femoral nerve block using ropivacaine 0.025%, 0.05% and 0.1%: effects on the rehabilitation programme following total knee arthroplasty: a pilot study. Anaesthesia. 2008 Sep;63(9):948-53. doi: 10.1111/j.1365-2044.2008.05538.x. Epub 2008 Jun 6. PMID 18540926
- [Background] de Leeuw MA, Dertinger JA, Hulshoff L, Hoeksema M, Perez RS, Zuurmond WW, de Lange JJ. The efficacy of levobupivacaine, ropivacaine, and bupivacaine for combined psoas compartment-sciatic nerve block in patients undergoing total hip arthroplasty. Pain Pract. 2008 Jul-Aug;8(4):241-7. doi: 10.1111/j.1533-2500.2008.00209.x. Epub 2008 May 23. PMID 18503623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-one patients signed an informed consent form. Eleven patients were excluded: six for inability to achieve <0.5mA quadriceps stimulation for lumbar plexus block placement and five for general anesthesia. After pharmacy randomization, 14 received ropivacaine 0.1% and 16 received ropivacaine 0.2%.
Groups:
- 0.2% Ropivacaine: 0.2% ropivacaine
  Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuous lumbar plexus catheters will be removed on post operative day (POD) 2.
- 0.1% Ropivacaine: 0.1% ropivacaine
  Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuous lumbar plexus catheters will be removed on post operative day (POD) 2.
Period: Overall Study
Arm/Group | 0.2% Ropivacaine | 0.1% Ropivacaine
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2% Ropivacaine | 0.1% Ropivacaine | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.8) | 56.1 (10.8) | 57.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Opiate Consumption Postoperatively
Description: Postoperative opiate consumption at 24 hours
Time Frame: 24 hours postoperatively
Population: Forty-one patients signed informed consent and underwent primary THA. Eleven patients were excluded: six for inability to achieve <0.5mA quadriceps stimulation for lumbar plexus block and five for general anesthesia. The study was completed after pharmacy randomization 30 patients: 16 in 0.2% and 14 in 0.1% group.
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | 0.2% Ropivacaine | 0.1% Ropivacaine
Number analyzed (Participants) | 16 | 14
mg | 8.21 [5.75 to 10.69] | 8.02 [6.02 to 10.02]

2. Secondary Outcome: Patient Satisfaction With Pain Control
Description: Patient satisfaction with pain control at 24 hours (0-10 scale). Patients' satisfaction was assessed using an 11-point numeric scale (0-10, 0 = unsatisfied and 10 = very satisfied). Scores at 24 hours were not averaged with any other scores.
Time Frame: 24 hours postoperatively
Population: Patient satisfaction with pain control at 24 hours.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- 0.1% Ropivacaine Infusion in Nerve Block Catheter: 0.1% ropivacaine
  Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuous lumbar plexus catheters will be removed on post operative day (POD) 2.
Arm/Group | 0.2% Ropivacaine | 0.1% Ropivacaine Infusion in Nerve Block Catheter
Number analyzed (Participants) | 16 | 14
units on a scale | 8 [7 to 9] | 9 [7 to 10]

3. Secondary Outcome: Numeric Rating Scale Pain Score With Movement at 24 Hours
Description: Numeric rating scale (NRS) pain score with movement were assessed at 24 hours. Pain scores were followed using an 11-point NRS (0 = no pain and 10 = worst imaginable pain). Scores at 24 hours were not averaged with any other scores.
Time Frame: 24 hours postoperatively
Population: NRS pain scores at 24 hours postoperatively at rest and in movement.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- 0.2% Ropivacaine Nerve Block (Standard of Care): 0.1% or 0.2% ropivacaine nerve blocks: Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuo
- 0.1% Ropivacaine Infusion in Nerve Block Catheter: 0.1% or 0.2% ropivacaine nerve blocks: Either 0.1% or 0.2% ropivacaine will be infused at 7 mL/hr through lumbar plexus nerve block catheter based upon randomization, and can then receive a 6 ml bolus of either 0.1% or 0.2% ropivacaine. Additional pain relief will be available by nurse administered boluses of additional local anesthetic (from their randomized infusion) with a maximum dose of an extra 3 ml per bolus and limited to one bolus per hour. This bolus of their randomized local anesthetic will remain available until the nerve catheters are removed. Nerve block infusion rates may be increased to 9 ml/h for patients with increased pain without increased motor blockade as determined by the acute interventional perioperative pain service (AIPPS) or decreased to 5 ml/h for patients with increased motor blockade or weakness from the peripheral nerve block as determined by the AIPPS .All continuous lumbar plexus catheters w
Arm/Group | 0.2% Ropivacaine Nerve Block (Standard of Care) | 0.1% Ropivacaine Infusion in Nerve Block Catheter
Number analyzed (Participants) | 16 | 14
units on a scale | 7 [4 to 9] | 7 [5 to 9]

4. Secondary Outcome: Number of Participants With Increased Infusion Rates
Description: Number of patients requiring increased infusion rates to 9 mL/hour to better optimize pain control.
Time Frame: Subjects will be followed postoperatively until postoperative day 2 (i.e. the discontinuation of the lumbar plexus catheters)
Population: The number of participants with requiring increased infusion rates.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2% Ropivacaine Nerve Block (Standard of Care) | 0.1% Ropivacaine Infusion in Nerve Block Catheter
Number analyzed (Participants) | 16 | 14
Participants | 4 | 3

5. Secondary Outcome: Number of Participants With Decreased Infusion Rates
Description: Number of patient requiring decreased infusion rates decreased to 5 mL/hour due to increased motor blockade.
Time Frame: as for outcome 4
Population: Number of patient requiring decreased infusion rates.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2% Ropivacaine Nerve Block (Standard of Care) | 0.1% Ropivacaine Infusion in Nerve Block Catheter
Number analyzed (Participants) | 16 | 14
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event were analyzed after lumbar plexus perineural catheter removal on POD2 as this was the end of the data collection period.
Arm/Group | 0.2% Ropivacaine | 0.1% Ropivacaine Infusion in Nerve Block Catheter
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No